CLINICAL TRIAL: NCT01790295
Title: Exploring the Potential of Dual Kinase JAK 1/2 Inhibitor Ruxolitinib (INC424) With Reduced Intensity Allogeneic Hematopoietic Cell Transplantation in Patients With Myelofibrosis
Brief Title: Ruxolitinib Prior to Transplant in Patients With Myelofibrosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: John Mascarenhas (Other)
Collaborators: Myeloproliferative Disorders-Research Consortium (Network); National Cancer Institute (NCI) (NIH); Incyte Corporation (Industry); Novartis (Industry)
Responsible Party: Sponsor-Investigator, John Mascarenhas, Associate Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 12-1809; MPD-RC 114
Record Dates: First submitted 2013-02-08; First posted 2013-02-13 (Estimated); Results first posted 2019-03-20 (Actual); Last update posted 2019-03-20 (Actual); Status verified 2019-02

CONDITIONS: Primary Myelofibrosis; Post Polycythemia Vera Myelofibrosis; Post Essential Thrombocythemia Myelofibrosis
Keywords: Myelofibrosis; Stem cell transplant; Ruxolitinib
MeSH Terms: conditions — Primary Myelofibrosis | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ruxolitinib Pre- Hematopoietic cell transplantation (HCT) (Experimental): Ruxolitinib (INC424) tablets will be started 62 days (day -67) prior to start of conditioning chemotherapy. The starting dose of Ruxolitinib will be determined according to baseline platelet count and will be modified according to platelet count at follow-up. The drug will be given in the maximum tolerated dose as defined in the protocol for 56 days, followed by 4 days of taper, and will be stopped completely at the planned start of conditioning therapy (starting on day -5) i.e. 5 days prior to stem cell infusion. The drug will be supplied as 5 mg tablets.
  Interventions: Drug: Ruxolitinib Pre- Hematopoietic cell transplantation (HCT)

INTERVENTIONS:
Drug: Ruxolitinib Pre- Hematopoietic cell transplantation (HCT) — Ruxolitinib (INC424) tablets will be started 60 days (day -65) prior to start of conditioning chemotherapy. The starting dose of Ruxolitinib will be determined according to baseline platelet count and will be modified according to platelet count at follow-up. The drug will be given in the maximum tolerated dose as defined in the protocol for 56 days, followed by 4 days of taper, and will be stopped completely at the planned start of conditioning therapy (starting on day -5) i.e. 5 days prior to stem cell infusion. The drug will be supplied as 5 mg tablets.
  Other Names: Ruxolitinib \Pre- Hematopoietic cell transplantation (HCT); INC424

SUMMARY:
The purpose of this study is to find out if giving the study drug Ruxolitinib (INC424) prior to a combination of other chemotherapeutic drugs (Fludarabine and Busulfan) before infusing another person's hematopoietic stem cells (bone marrow transplantation) will be successful in people who have advanced primary myelofibrosis (PMF), post-polycythemia vera myelofibrosis (PPV-MF) or post-essential thrombocythemia myelofibrosis (PET-MF), collectively known as myelofibrosis (MF). MF is a disorder in which bone marrow tissue develops in abnormal sites because the bone marrow itself undergoes fibrosis or scarring. This study plans to evaluate whether adding the drug Ruxolitinib will further aid in reducing pre-transplant spleen size, improve physical performance levels and reduce adverse events (side effects) related to the transplant. Ruxolitinib is a drug that is approved by the FDA for the treatment of patients with advanced forms of myelofibrosis. Using Ruxolitinib prior to stem cell transplantation is experimental.

DETAILED DESCRIPTION:
A two- stage Simon Phase II study will be conducted in each of two groups of patients: related and unrelated donor transplants. In each donor transplant group, the first stage of this design will include 11 patients evaluated for death or graft failure by 100 days post-transplant. In each stratum, we will enroll additional patients (up to 20%) of stratum total to take into account exclusions due to donor failure (such as donor deemed unsuitable for stem cell donation due to medical or other reasons) only. Those patients who have toxicities related to Ruxolitinib and not been able to reach HCT due to these toxicities will be included in the estimation of overall failure rates. Only those patients who are excluded based on donor related issues without any regimen related complications will be excluded from the estimation of failure rates. However, all data on these patients will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of primary myelofibrosis according to WHO criteria or post PV myelofibrosis or post ET myelofibrosis as per IWG-MRT criteria
* Age 18-70 years
* Intermediate-2/ high-risk disease as per Dynamic IPSS (DIPSS) criteria OR Intermediate-1 risk disease with one of the following additional unfavorable features known to impact the survival adversely

  1. Red cell transfusion dependency
  2. Unfavorable Karyotype
  3. Platelet count <100 x 109/l
* Blasts in the PB and BM ≤10% prior to study enrollment
* Availability of a suitable matched related (6/6 or 5/6) or unrelated donor (10/10 or 9/10 antigen or allele matched).
* Able to give informed written consent
* ECOG Performance status of 0-2.
* Life expectancy >3 months
* Off all MF-directed therapy including investigational agents for at least 2 weeks prior to study enrollment and recovered from all toxicities*
* Adequate organ function

  * Adequate renal function - creatinine <1.5 x IULN
  * Adequate hepatic function - AST/ALT <2.5 x IULN, Total Bilirubin <1.5 x IULN
  * Adequate hematopoietic function - Platelet ≥50 x 109/l and ANC ≥1.0 x 109/l
  * LVEF >40% (MUGA or echocardiogram) Normal per Institutional standard
  * Adequate pulmonary function with DLCO >50%

    * A patient who has been on stable dose of Ruxolitinib and has received ruxolitinib ≤6 months prior to the study entry will be considered potentially eligible for the study with the caveat that there is no evidence of loss of response (>5cm increase in spleen size from the nadir).

Exclusion Criteria:

* Any previous JAK2 inhibitor treatment prior to study enrollment, with the exception of Ruxolitinib
* Hypersensitivity to JAK inhibitor
* Clinical or laboratory evidence of cirrhosis
* Prior allogeneic transplant for any hematopoietic disorder
* >20% blast in the PB or BM prior to HCT or had leukemic transformation (>20% blasts in PB or BM any time prior to HCT)
* Syngeneic donor
* Cord Blood transplant
* Active uncontrolled infection
* H/o another malignancy within 5-years of date of HCT except h/o basal cell or squamous cell carcinoma of skin or PV or ET
* Known HIV positive
* Pregnancy at the time of BMT
* Any other concurrent illness which in investigator's opinion puts the patient at excessive risk of treatment related toxicities
* Unable to give informed consent
* Active infection with hepatitis A,B or C virus
* Subjects who require therapy with a strong CYP3A4 inhibitor prior to enrollment to this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-11; Primary Completion 2017-10-26 (Actual); Study Completion 2017-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Mascarenhas, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Vikas Gupta, MD, FRCP, FRCPath, Study Chair — University of Toronto; Adam Mead, MD, Study Chair — University of Oxford, John Radcliffe Hospital
Locations (8):
- United States (6):
  - Emory Hospital, Atlanta, Georgia
  - Northwestern University, Robert h. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - University of Kansas Cancer Center, Westwood, Kansas
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
- Princess Margaret Cancer Centre, University of Toronto, Toronto, Canada
- University of Oxford, Oxford, United Kingdom

REFERENCES:
- [Derived] Gupta V, Kosiorek HE, Mead A, Klisovic RB, Galvin JP, Berenzon D, Yacoub A, Viswabandya A, Mesa RA, Goldberg J, Price L, Salama ME, Weinberg RS, Rampal R, Farnoud N, Dueck AC, Mascarenhas JO, Hoffman R. Ruxolitinib Therapy Followed by Reduced-Intensity Conditioning for Hematopoietic Cell Transplantation for Myelofibrosis: Myeloproliferative Disorders Research Consortium 114 Study. Biol Blood Marrow Transplant. 2019 Feb;25(2):256-264. doi: 10.1016/j.bbmt.2018.09.001. Epub 2018 Sep 8. PMID 30205231

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in February 2013, with first enrollment in November 2013.
Groups:
- Ruxolitinib Pre- Hematopoietic Cell Transplantation (HCT): Ruxolitinib Pre- Hematopoietic cell transplantation (HCT) in Patients With Myelofibrosis.
  Ruxolitinib (INC424) tablets started 60 days (day -65) prior to start of conditioning chemotherapy. The starting dose of Ruxolitinib was determined according to baseline platelet count and modified according to platelet count at follow-up. The drug was given in the maximum tolerated dose as defined in the protocol for 56 days, followed by 4 days of taper, and stopped completely at the planned start of conditioning therapy (starting on day -5) i.e. 5 days prior to stem cell infusion. The drug was supplied as 5 mg tablets.
Period: Overall Study
Arm/Group | Ruxolitinib Pre- Hematopoietic Cell Transplantation (HCT)
Started | 21
Completed | 10
Not Completed | 11
Not completed — Adverse Event | 1
Not completed — Death | 4
Not completed — Lack of Efficacy | 2
Not completed — Study closure | 4

BASELINE CHARACTERISTICS:
Groups:
- Ruxolitinib Pre- Hematopoietic Cell Transplantation (HCT): Ruxolitinib Pre- Hematopoietic cell transplantation (HCT) in Patients With Myelofibrosis
  Ruxolitinib (INC424) tablets started 60 days (day -65) prior to start of conditioning chemotherapy. The starting dose of Ruxolitinib was determined according to baseline platelet count and modified according to platelet count at follow-up. The drug was given in the maximum tolerated dose as defined in the protocol for 56 days, followed by 4 days of taper, and stopped completely at the planned start of conditioning therapy (starting on day -5) i.e. 5 days prior to stem cell infusion. The drug was supplied as 5 mg tablets.
Arm/Group | Ruxolitinib Pre- Hematopoietic Cell Transplantation (HCT)
Number analyzed (Participants) | 21
Age, Continuous [Median (Full Range); unit: years] | 59 [39 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0
Diagnosis [Count of Participants; unit: Participants] — Primary Myelofibrosis Post Polycythemia Vera (Post-PV) Myelofibrosis Post Essential Thrombocythemia (Post-ET) Myelofibrosis
  Participants
    Primary myelofibrosis | 10
    Post-PV myelofibrosis | 3
    Post-ET myelofibrosis | 8
Donor type [Count of Participants; unit: Participants]
  Related donor | 7
  Unrelated donor | 14
ECOG status [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) measures level of functioning in terms of daily living abilities:
  The ECOG measures level of functioning in terms of daily living abilities:
  0-Fully active, able to carry on all pre-disease performance without restriction
  1-Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, eg.light house work
  Participants
    0 | 9
    1 | 12

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With 100-day Survival Without Graft Failure
Description: The feasibility of combining Ruxolitinib (INC424) with a Reduced intensity conditioning (RIC) regimen likely to produce success post transplantation, success being defined as patient being alive, and without graft failure at day 100-post allogeneic stem cell transplantation (in patients who receive (a) related donor transplant and in those who receive (b) an unrelated donor transplant.
Time Frame: Day 100-post allogeneic stem cell transplantation
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib Pre- Hematopoietic Cell Transplantation (HCT)
Number analyzed (Participants) | 21
percentage of participants | 74 [48 to 88]

2. Secondary Outcome: Time to Neutrophil Recovery
Description: Neutrophil recovery will be defined as first of the three consecutive days with neutrophil count ≥0.5 x 109/l.
Time Frame: up to 4 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ruxolitinib Pre- Hematopoietic Cell Transplantation (HCT)
Number analyzed (Participants) | 21
days | 23 [13 to 31]

3. Secondary Outcome: Platelet Recovery
Description: Platelet recovery will be defined as first of the 7 days with platelet count ≥20 x 109/l, without platelet transfusion support and both maintained for 30 days without transfusion support or myeloid cytokine support.
Time Frame: up to 4 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Ruxolitinib Pre- Hematopoietic Cell Transplantation (HCT)
Number analyzed (Participants) | 21
days | 30 [18 to 57]

4. Secondary Outcome: Percent of Participants With Non-relapse Mortality (NRM)
Description: NRM will be defined as death in first 30 days due to any cause, and subsequently death due to any cause without the recurrence or progression of myelofibrosis. Cumulative incidence of NRM will be calculated taking relapse/progression as competing event.
Time Frame: 100 days
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib Pre- Hematopoietic Cell Transplantation (HCT)
Number analyzed (Participants) | 21
percentage of participants | 16 [5 to 46]

5. Secondary Outcome: Percent of Participants With Non-relapse Mortality (NRM)
Description: as for outcome 4
Time Frame: 1-year post transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib Pre- Hematopoietic Cell Transplantation (HCT)
Number analyzed (Participants) | 21
percentage of participants | 28 [13 to 61]

6. Secondary Outcome: Percent of Participants With Graft Versus Host Disease (GvHD)
Description: Acute and chronic GvHD. GvHD is a potentially serious complication of allogeneic stem cell transplantation.
  Stage Skin Liver (bilirubin) Gut (stool output/day)
  0 No GVHD rash < 2 mg/dl < 500 ml/day or persistent nausea.
  1. Maculopapular rash< 25% body surface area (BSA) 2-3 mg/dl 500-999 ml/day
  2. Maculopapular rash 25 - 50% BSA 3.1-6 mg/dl 1000-1500 ml/day
  3. Maculopapular rash > 50% BSA 6.1-15 mg/dl Adult: >1500 ml/day
  4. Generalized erythroderma plus bullous formation >15 mg/dl Severe abdominal pain with or without ileus Grade I Stage 1-2 None None II Stage 3 or Stage 1 or Stage 1 III - Stage 2-3 or Stage 2-4 IV Stage 4 or Stage 4 -
Time Frame: 1-year post transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Ruxolitinib Pre- Hematopoietic Cell Transplantation (HCT)
Number analyzed (Participants) | 21
percentage of participants
  Acute GvHD (Grade 1/2) | 48 [29 to 79]
  Acute GvHD (Grade 3) | 16 [5 to 46]
  Chronic GvHD (Mild) | 51 [31 to 86]
  Chronic (Moderate) | 25 [9 to 72]

7. Secondary Outcome: Chimerism Studies
Description: Will check percentage of donor versus recipient blood cells to determine efficacy of donor engraftment
Time Frame: 30 days post transplant
Population: This data was not collected because the study ended early.
Arm/Group | Ruxolitinib Pre- Hematopoietic Cell Transplantation (HCT)
Number analyzed (Participants) | 0

8. Secondary Outcome: Chimerism Studies
Description: Will check percentage of donor versus recipient blood cells to determine efficacy of donor engraftment
Time Frame: 60 days post transplant
Population: This data was not collected because the study ended early.
Groups:
- Ruxolitinib Pre- Hematopoietic Cell Transplantation (HCT): Ruxolitinib Pre- Hematopoietic cell transplantation (HCT) in Patients With Myelofibrosis
Arm/Group | Ruxolitinib Pre- Hematopoietic Cell Transplantation (HCT)
Number analyzed (Participants) | 0

9. Secondary Outcome: Chimerism Studies
Description: Will check percentage of donor versus recipient blood cells to determine efficacy of donor engraftment
Time Frame: 100 days post transplant
Population: This data was not collected because the study ended early.
Arm/Group | Ruxolitinib Pre- Hematopoietic Cell Transplantation (HCT)
Number analyzed (Participants) | 0

10. Secondary Outcome: Number of Participants With Remission Status According to IWG-MRT Criteria
Description: Remission status according to International Working Group for Myelofibrosis Research and Treatment (IWG-MRT) criteria
  Remission defined as:
  Bone marrow:* Age-adjusted normocellularity; <5% blasts; ≤grade 1 MF and Peripheral blood: Hemoglobin ≥100 g/L and <UNL; neutrophil count ≥ 1 × 109/L and <UNL; Platelet count ≥100 × 109/L and <UNL; <2% immature myeloid cells and Clinical: Resolution of disease symptoms; spleen and liver not palpable; no evidence of extramedullary hematopoiesis (EMH)
Time Frame: Day 100 post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib Pre- Hematopoietic Cell Transplantation (HCT)
Number analyzed (Participants) | 21
Participants | 20

11. Secondary Outcome: Number of Participants With Remission Status at 6 Months Post Transplant
Description: Remission defined as:
  Bone marrow:* Age-adjusted normocellularity; <5% blasts; ≤grade 1 MF† and Peripheral blood: Hemoglobin ≥100 g/L and <UNL; neutrophil count ≥ 1 × 109/L and <UNL; Platelet count ≥100 × 109/L and <UNL; <2% immature myeloid cells‡ and Clinical: Resolution of disease symptoms; spleen and liver not palpable; no evidence of EMH
Time Frame: 6 months post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib Pre- Hematopoietic Cell Transplantation (HCT)
Number analyzed (Participants) | 21
Participants | 17

12. Secondary Outcome: Number of Participants With Remission Status at 12 Months Post Transplant
Description: as for outcome 11
Time Frame: 12 months post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib Pre- Hematopoietic Cell Transplantation (HCT)
Number analyzed (Participants) | 21
Participants | 14

13. Secondary Outcome: Number of Participants With Relapse/Progression (Defined as Per IWG-MRT Criteria)
Description: Relapse/progression defined as:
  Peripheral blood: Hemoglobin ≥100 g/L and <UNL; neutrophil count ≥1 × 109/L and <UNL; platelet count ≥100 × 109/L and <UNL; <2% immature myeloid cells‡ and Clinical: Resolution of disease symptoms; spleen and liver not palpable; no evidence of EMH or Bone marrow:* Age-adjusted normocellularity; <5% blasts; ≤grade 1 MF†, and peripheral blood: Hemoglobin ≥85 but <100 g/L and <UNL; neutrophil count ≥1 × 109/L and <UNL; platelet count ≥50, but <100 × 109/L and <UNL; <2% immature myeloid cells‡ and Clinical: Resolution of disease symptoms; spleen and liver not palpable; no evidence of EMH
Time Frame: 1-year post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib Pre- Hematopoietic Cell Transplantation (HCT)
Number analyzed (Participants) | 21
Participants | 7

14. Secondary Outcome: Number of Participants With Progression-free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 1-year post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib Pre- Hematopoietic Cell Transplantation (HCT)
Number analyzed (Participants) | 21
Participants | 11

15. Secondary Outcome: Number of Overall Survival
Time Frame: 1-year post transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Ruxolitinib Pre- Hematopoietic Cell Transplantation (HCT)
Number analyzed (Participants) | 21
Participants | 15

16. Secondary Outcome: Mean Change in the Brief Fatigue Inventory Score
Description: Mean change in the Brief Fatigue Inventory score (BFI) from baseline to 48 months to assess impact of allogeneic stem cell transplant on myelofibrosis associated symptoms and overall quality of life. The BFI is a 9 item scored from 0 (no fatigue) -10 (as bad as you can imagine), items are averaged with total score from 0-10, with higher score indicating more fatigue.
Time Frame: baseline and 48 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Ruxolitinib Pre- Hematopoietic Cell Transplantation (HCT)
Number analyzed (Participants) | 21
score on a scale | 1.7 [0.25 to 3.08]

17. Secondary Outcome: Expression Profiling and Measurements of Cytokines Prior to Start of Ruxolitinib, Prior to Start of Chemotherapy for Conditioning
Time Frame: 30 days post transplant
Population: This data was not collected because the study ended early.
Arm/Group | Ruxolitinib Pre- Hematopoietic Cell Transplantation (HCT)
Number analyzed (Participants) | 0

18. Secondary Outcome: Expression Profiling and Measurements of Cytokines Prior to Start of Ruxolitinib, Prior to Start of Chemotherapy for Conditioning
Time Frame: 100 days post transplant
Population: This data was not collected because the study ended early.
Arm/Group | Ruxolitinib Pre- Hematopoietic Cell Transplantation (HCT)
Number analyzed (Participants) | 0

19. Secondary Outcome: Association of Cytokines Levels With Acute and Chronic GvHD
Time Frame: 30 days post transplant
Population: This data was not collected because the study ended early.
Arm/Group | Ruxolitinib Pre- Hematopoietic Cell Transplantation (HCT)
Number analyzed (Participants) | 0

20. Secondary Outcome: Association of Cytokines Levels With Acute and Chronic GvHD
Time Frame: 100 days post transplant
Population: This data was not collected because the study ended early.
Arm/Group | Ruxolitinib Pre- Hematopoietic Cell Transplantation (HCT)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: up to 4 years
Arm/Group | Ruxolitinib Pre- Hematopoietic Cell Transplantation (HCT)
All-Cause Mortality (participants affected / at risk) | 4/21
Serious Adverse Events (participants affected / at risk) | 13/21
Other Adverse Events (participants affected / at risk) | 20/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib Pre- Hematopoietic Cell Transplantation (HCT) (N=21)
Drug-induced hyperglycemia (Endocrine disorders) | 1
Diverticulitis NOS (Gastrointestinal disorders) | 1
Nausea post chemotherapy (Gastrointestinal disorders) | 1
Death sudden (General disorders) | 1
Neutropenic fever (General disorders) | 1
Pneumonia (Infections and infestations) | 4
Sepsis (Infections and infestations) | 3
Graft failure (Injury, poisoning and procedural complications) | 4
Elevated liver enzyme levels (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Intracranial hemorrhage (Nervous system disorders) | 1
Spinal epidural hematoma (Nervous system disorders) | 1
Acute renal failure (Renal and urinary disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Disease Progression (General disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ruxolitinib Pre- Hematopoietic Cell Transplantation (HCT) (N=21)
Abdominal pain (Gastrointestinal disorders) | 9
Activated partial thromboplastin time (Investigations) | 5
Acute kidney injury (Renal and urinary disorders) | 4
Acute myeloid leukemia (Blood and lymphatic system disorders) | 1
Acute renal failure (Renal and urinary disorders) | 1
Agitation (Nervous system disorders) | 1
Alanine aminotransferase increased (Investigations) | 7
Alkaline phosphatase increased (Investigations) | 7
Allergic rash (Skin and subcutaneous tissue disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3
Alloimmunization (Immune system disorders) | 1
Anal hemorrhage (Gastrointestinal disorders) | 3
Anemia (Blood and lymphatic system disorders) | 13
Ankle edema (Musculoskeletal and connective tissue disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 7
Anxiety (Psychiatric disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Back pain (without radiation) (Musculoskeletal and connective tissue disorders) | 6
Bloating (Gastrointestinal disorders) | 5
Blood bilirubin increased (Investigations) | 5
Blurred vision (Eye disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Bronchospasm (Immune system disorders) | 1
Bruising (Skin and subcutaneous tissue disorders) | 5
Burning from urination (Renal and urinary disorders) | 1
Burning sensation (Nervous system disorders) | 1
C.difficile diarrhea (Gastrointestinal disorders) | 1
CMV infection (Infections and infestations) | 1
Cardiac neoplasm unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cardiomyopathy (Cardiac disorders) | 1
Cataract (Eye disorders) | 1
Catheter site erythema (General disorders) | 1
Chest congestion (Respiratory, thoracic and mediastinal disorders) | 1
Chest pain - cardiac (Cardiac disorders) | 1
Chills (General disorders) | 6
Chronic kidney disease (Renal and urinary disorders) | 1
Clostridium difficile test positive (Infections and infestations) | 1
Confusion (Nervous system disorders) | 2
Confusion (Psychiatric disorders) | 2
Conjunctivitis (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Contusion (Vascular disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Creatinine increased (Investigations) | 4
Cytokine release syndrome (Immune system disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Delirium (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 4
Diaphoresis (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 11
Dizziness (Nervous system disorders) | 8
Double vision (Eye disorders) | 1
Drug-induced liver disease (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Dry mouth (Gastrointestinal disorders) | 6
Dry skin (Skin and subcutaneous tissue disorders) | 6
Dysgeusia (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 5
Dysphagia (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10
Ear pain (Ear and labyrinth disorders) | 2
Edema extremities (General disorders) | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
Erythema (Skin and subcutaneous tissue disorders) | 3
Facial swelling (Skin and subcutaneous tissue disorders) | 1
Fall (Injury, poisoning and procedural complications) | 2
Fatigue (General disorders) | 8
Febrile neutropenia (Blood and lymphatic system disorders) | 6
Fecal incontinence (Gastrointestinal disorders) | 2
Fever (General disorders) | 8
Fibrinogen decreased (Investigations) | 1
Flatulence (Gastrointestinal disorders) | 2
Folliculitis (Skin and subcutaneous tissue disorders) | 2
Foot injury (Injury, poisoning and procedural complications) | 1
GGT Increased (Metabolism and nutrition disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5
Gout (Metabolism and nutrition disorders) | 1
Gynecomastia (Reproductive system and breast disorders) | 1
HSV infection (Infections and infestations) | 1
Headache (Nervous system disorders) | 8
Hearing impaired (Ear and labyrinth disorders) | 1
Hematoma (Vascular disorders) | 1
Hematuria (Renal and urinary disorders) | 2
Hemoglobin decreased (Investigations) | 1
Hemolysis (Blood and lymphatic system disorders) | 1
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 9
Hyperkalemia (Metabolism and nutrition disorders) | 8
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypertension (Metabolism and nutrition disorders) | 6
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 8
Hypocalcemia (Metabolism and nutrition disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 10
Hyponatremia (Metabolism and nutrition disorders) | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 5
Hypotension (Vascular disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
INR increased (Investigations) | 5
Increased TSH (Investigations) | 1
Infusion site cellulitis (Infections and infestations) | 1
Insomnia (Nervous system disorders) | 2
Insufficiency adrenal (Endocrine disorders) | 1
Iron deficiency anemia (Blood and lymphatic system disorders) | 1
Irritation lips (Gastrointestinal disorders) | 1
Itching (Skin and subcutaneous tissue disorders) | 1
Laboratory test abnormal (Investigations) | 1
Left lower quadrant pain (Gastrointestinal disorders) | 1
Lethargy (General disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Lightheadedness (Vascular disorders) | 1
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1
Lymphocyte count decreased (Investigations) | 5
Lymphocyte count increased (Investigations) | 1
Maculopapular rash (Skin and subcutaneous tissue disorders) | 3
Malaise (General disorders) | 2
Middle ear inflammation (Ear and labyrinth disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 8
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Nausea (Gastrointestinal disorders) | 14
Nausea and vomiting (Gastrointestinal disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Neutrophil count decreased (Investigations) | 9
Night blindness (Eye disorders) | 11
Night sweats (General disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Open wound of foot except toe(s) alone (Injury, poisoning and procedural complications) | 1
Oral hemorrhage (Gastrointestinal disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
Pain (General disorders) | 4
Painful urination (Renal and urinary disorders) | 1
Palpitations (Cardiac disorders) | 1
Paraplegia (Nervous system disorders) | 1
Perianal pain (Gastrointestinal disorders) | 1
Periocular rash (Skin and subcutaneous tissue disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Petechiae (Blood and lymphatic system disorders) | 4
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1
Plasma creatinine increased (Investigations) | 1
Platelet count decreased (Investigations) | 10
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Polymyalgia rheumatica (Immune system disorders) | 1
Post procedural discomfort (General disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Pressure sore (Skin and subcutaneous tissue disorders) | 1
Presyncope (Cardiac disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5
Pseudogout (Musculoskeletal and connective tissue disorders) | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 1
Renal calculi (Renal and urinary disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory syncytial virus infection (Infections and infestations) | 12
Rigors (General disorders) | 1
Scleral hemorrhage (Eye disorders) | 2
Sepsis (Infections and infestations) | 1
Sinus tachycardia (Cardiac disorders) | 4
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1
Skin desquamation (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin infection (Infections and infestations) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnea (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 2
Sore throat (Gastrointestinal disorders) | 4
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4
Syncope (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Tooth pain (Gastrointestinal disorders) | 1
Tremor (Nervous system disorders) | 2
Upper respiratory tract infection bacterial (Infections and infestations) | 3
Urinary incontinence (Nervous system disorders) | 2
Urinary hesitancy (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 2
Urinary tract infection (Infections and infestations) | 2
Urticaria (Immune system disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Weakness (General disorders) | 1
Weight gain (Investigations) | 1
Weight loss (Investigations) | 5
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4
White blood cell decreased (Investigations) | 9
Aspartate aminotransferase increased (Investigations) | 8
Autoimmune hemolytic anemia (Blood and lymphatic system disorders) | 1
Edema periorbital (Skin and subcutaneous tissue disorders) | 1
Edematous weight gain (General disorders) | 1
Hypoalbuminemia (Hepatobiliary disorders) | 8
Macular Rash (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 4
Syncope (Nervous system disorders) | 2
White blood cell count increased (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2016-08-08): https://cdn.clinicaltrials.gov/large-docs/95/NCT01790295/Prot_SAP_ICF_000.pdf